CLINICAL TRIAL: NCT03703570
Title: A Phase 2b Study of KW-6356 in Subjects With Parkinson's Disease on Treatment With Levodopa-containing Preparations
Brief Title: A Study of KW-6356 in Patients With Parkinson's Disease on Treatment With Levodopa-containing Preparations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6356-003
Record Dates: First submitted 2018-10-05; First posted 2018-10-12 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: An interventional, multicenter, randomized, double-blind, placebo-controlled, parallel-group trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KW-6356 Low Dose (Experimental): Oral administration
  Interventions: Drug: KW-6356
- KW-6356 High Dose (Experimental): Oral administration
  Interventions: Drug: KW-6356
- placebo (Placebo Comparator): Oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KW-6356 — Oral administration
  Arms: KW-6356 High Dose; KW-6356 Low Dose
Drug: Placebo — Oral administration
  Arms: placebo

SUMMARY:
The primary objective of this study is to determine the recommended dose and evaluate the effect of KW-6356 on motor symptoms in Parkinson's disease and the primary endpoint is the change from baseline in Movement disorder society-unified Parkinson's disease rating scale(MDS-UPDRS) partIII score between KW-6356 and placebo in patients with Parkinson's disease on treatment with Levodopa-containing preparations as an adjunctive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject fulfills the UK Parkinson's Disease Society brain bank clinical diagnostic criteria.
* Parkinson's disease patients in Stages 2 to 4 on the Modified Hoehn and Yahr Scale. (mH&Y, Evaluation at ON state for patients who experience Wearing-off phenomenon)
* MDS-UPDRS partIII score of >= 15. (Evaluation at ON state)
* Subject who are responsive to levodopa/DCI (carbidopa or benserazide) combination therapy and who have been on the therapy for 6 months or longer without interruption at enrollment.
* Subject who have not started any new antiparkinsonian drugs and have been on a stable regimen of antiparkinsonian drugs in the 3 months before enrollment.

Exclusion Criteria:

* Use of any CYP3A4/5-related drugs within 2 weeks prior to enrollment.
* Use of any of the following drugs within 3 months (or 6 month in case of depot preparations) prior to enrollment; Antipsychotics, tiapride, metoclopramide, amoxapine, reserpine, tetrabenazine, methyldopa, papaverine, Levodopa/carbidopa intestinal gel and apomorphine hydrochloride injection
* Treatment by transcranial magnetic stimulation (TMS) within 6 months prior to enrollment.
* Neurosurgical operation for Parkinson's disease. (stereotactic surgery, deep brain stimulation or gamma knife)
* Subject who have received administration of adenosine A2A receptor antagonist.
* Either of the following criteria consecutively at screening and enrollment; Resting Pulse > 100 bpm Resting systolic blood pressure > 140 mmHg, or diastolic blood pressure > 90 mmHg
* Significant dementia or a Mini-Mental State Examination (MMSE) score of =< 23.
* Subject has a history or evidence of suicidal ideation (severity of 4 or 5) or any suicidal behavior based on an assessment with the Columbia-Suicide Severity Rating Scale (C-SSRS) at baseline.
* Anyone otherwise considered unsuitable for the study by the investigator or subinvestigator including those who are unable to communicate or to cooperate with the investigator or subinvestigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Movement disorder society-unified Parkinson's disease rating scale(MDS-UPDRS) part III score | Up to 26 weeks after dosing
  MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The scales are now titled; (Part I) nonmotor experiences of daily living (13 items), (Part II) motor experiences of daily living (13 items), (Part III) motor examination (18 items), and (Part IV) motor complications (six items). Each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.
  The total score is the sum of the subscale scores for Parts III and ranges from 0 (no disability) to 136 (total dependence).

SECONDARY OUTCOMES:
Change from baseline in the total hours of awake time per day spent in the OFF state. (total hours per day spent in the OFF state) | Up to 26 weeks after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Iwamizawa Neurology Clinic, Iwamizawa, Hokkaido, Japan